CLINICAL TRIAL: NCT04826653
Title: Influence of Timing Suture Removal on Root Coverage Procedures: a Randomized Prospective Clinical Trial
Brief Title: Timing Suture Removal on Root Coverage Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Clinical Instructor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PER-ECL-2019-02
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Gingival Recession; Suture; Root Coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Timing suture removal_1 week (Experimental)
  Interventions: Other: Suture removal
- Timing suture removal_2 weeks (Experimental)
  Interventions: Other: Suture removal
- Timing suture removal_3 weeks (Experimental)
  Interventions: Other: Suture removal

INTERVENTIONS:
Other: Suture removal — Suture removal after coronally advanced flap plus a connective tissue graft

SUMMARY:
Gingival recession is defined as the displacement of the soft tissue margin apical to the cemento-enamel junction with exposure of the root surface. It affects a broad population with presence of periodontal disease as well as periodontally healthy individuals. The occurrence of gingival recessions is age-dependent and their development begins relatively early in life. For instance, gingival recessions were noticed in more than 60% of Norwegian 20-year-olds and in more than 90% of the older population. Similar findings were reported in Brazilian and French population. In populations deprived of dental care, the occurrence of gingival recessions was even higher.

Many factors have been implicated in the etiology of gingival recession, including plaque, position of the tooth in the arch and improper toothbrushing. It is difficult to see a single cause for the development of labial gingival recession.

It has been demonstrated in several investigations that if left untreated, the probability of progression of the recession is high even with good oral hygiene. The indications for treatment of gingival recession are: esthetics, dental hypersensitivity, and the prevention of caries as well as further progression of the recession. Therapeutic options for recessions have been well documented with a high degree of success. Their ultimate goal is the location of the gingival margin coronal to the CEJ, with minimal probing depth and a pleasant soft tissue integration with the adjacent teeth.

With such a prevalent condition, it becomes critical to discriminate when to treat these lesions and which are the anatomical and surgical characteristics that are going to determine the amount of root coverage.

Regarding surgical characteristics, it has been demonstrated that the accomplishment of complete root coverage may be prejudiced by the post-surgical position of the gingival margin (the more coronal to the CEJ the greater the chance to achieve root coverage). The same author conducted a randomized clinical trial showing that the higher the flap tension, the lower the recession reduction. Another surgical factor affecting root coverage may be the use of microsurgical approaches by the use of smaller diameter sutures. According to a recently published systematic review, early suture removal (less than 10 days) can negatively affect root coverage outcome.

The healing process after pedicle graft was investigated in an animal model study. The healing was divided into four different stages, the adaption stage (0-4 days), the proliferation stage (4-21 days), the attachment stage (27-28 days) and the maturation stage (1-6 months). During the proliferation stage, connective tissue invades the fibrin layer from the basal level of the flap, and after 6-10 days a layer of fibroblasts is seen in apposition to the root surface. These cells are believed to differentiate into cementoblasts at a later stage of healing. At the end of the proliferation stage, thin collagen fibers are formed adjacent to the root surface, but a fibrous union between the connective tissue and the root has not been observed. It seems logical that stabilizing the flap with sutures for a prolonged period of time during the proliferation phase would help maintain the gingival margin on a more coronal position postoperatively. On the other hand, the longer the sutures remain postoperatively, the greater the chances of plaque accumulation and inflammation affecting negatively to root coverage.

The systematic review by Tatakis and Chambrone included 17 randomized clinical trials that provided an overall data of 325 single recession defects that were treated by coronally advanced flap. While they investigated time of suture removal, the studies included in this study did not account for this variable, thus leading to some bias. Moreover, different suture materials, type of suturing technique may also play an important role in the healing process. Therefore, the aim of this study is to evaluate the clinical outcome of timing suture removal regarding root coverage on coronally advanced flap.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* periodontally and systemically healthy
* presence of at least two consecutive Cairo type I (RT1) gingival recession defects
* recession >2mm in depth at the buccal aspect
* full-mouth plaque and bleeding score ≤20%
* no previous periodontal surgery; presence of identifiable cemento-enamel junction (CEJ) (a step 1mm at the CEJ and/or presence of root abrasion, but with identifiable CEJ, will be accepted).

Exclusion Criteria:

* smokers >10 cigarettes a day
* contraindications for periodontal surgery
* medications known to affect the gingiva or interfere with wound healing
* pregnancy and lactating females
* active orthodontic therapy
* caries or restorations in the area to be treated.
* Patients unable to follow post-surgical medication instructions adequately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Mean Root Coverage (MRC) in percentage (%) | 3- and 6-months post-surgery
  the average improvement in millimeters of the recession depth will be calculated as a percentage

SECONDARY OUTCOMES:
Complete root coverage (CRC) | 3- and 6-months post-surgery
Change in Keratinized Tissue Width (KT) at 3- and 6-months post-surgery. | 3- and 6-months post-surgery
Change in gingival thickness (GT) at 3- and 6-months post-surgery | 3- and 6-months post-surgery
Pain and discomfort of the suture of the grafted area. | 3- and 6-months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- International University of Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blasi G, Maury L, Lapedra A, Vilarrasa J, Monje A, Nart J. Suture Removal Timing and its Effect on Root Coverage: A Randomized Clinical Trial. Int J Periodontics Restorative Dent. 2025 Mar 4;0(0):1-26. doi: 10.11607/prd.7525. Online ahead of print. PMID 40036297